CLINICAL TRIAL: NCT01419834
Title: Phase I Study of Humanized 3F8 Monoclonal Antibody (Hu3F8) in Patients With High-Risk Neuroblastoma and GD2-Positive Tumors
Brief Title: Humanized 3F8 Monoclonal Antibody (Hu3F8) in Patients With High-Risk Neuroblastoma and GD2-Positive Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Band of Parents (Unknown); Y-mAbs Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-009
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Neuroblastoma
Keywords: CNS; Brain; MAB 3F8; Hu3F8; 11-009
MeSH Terms: conditions — Neuroblastoma | interventions — humanized 3F8 anti-GD2 monoclonal antibody

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Humanized 3F8 Monoclonal Antibody (Hu3F8) (Experimental): This phase I single arm trial assesses the toxicity of escalating doses of hu3F8.
  Interventions: Biological: Humanized 3F8 Monoclonal Antibody (Hu3F8)

INTERVENTIONS:
Biological: Humanized 3F8 Monoclonal Antibody (Hu3F8) — Hu3F8 is infused IV over ~30 minutes

SUMMARY:
The purpose of this study is to find out if "humanized 3F8" (Hu3F8) is safe for treating neuroblastoma and other cancers. A phase 1 study means the investigators are trying to find out what side effects happen when higher and higher doses of a drug are used.

The investigators want to find out what effects, good and/or bad, Hu3F8 has on cancer. The amount of Hu3F8 that patients gets will depend on when they start treatment on this study. The investigators also want to find out more about how Hu3F8 works and how effective it is in attacking the disease. Hu3F8 is an experimental drug, which means it has not yet been approved by the FDA for the treatment of this disease.

DETAILED DESCRIPTION:
Patients can be treated on 2 different schedules:

For patients following a 2 doses/cycle schedule (patients who were enrolled and started treatment prior to Amendment A(8)), one cycle has 2 days of intravenous hu3F8 treatment, given approximately 7 days apart.

For patients following a 3 doses/cycle schedule, one cycle has 3 days of intravenous hu3F8 treatment, given on days 1, 3 and 5. After Cycle 1, patients may receive treatment on a modified schedule of 3 days of intravenous hu3F8 over 10 days, as needed. To limit side-effects, patients receive analgesics and antihistamines as premedications. Cycles are 21 days and can be repeated up to a total of 12 cycles, see section 9.1 for details. Evaluations before, during and after treatment are summarized in Tables 4A and B. In addition, to further study the side effect of pain, patients will be asked to assess their pain on the days of treatment with hu3F8 at 3 different time points: (a) prior to commencement of hu3F8, (b) at least once during the acute pain episode when rescue pain medication doses are usually required and (c) prior to discharge from the Pediatric Day Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have either (1) a diagnosis of NB as defined by international criteria,56 i.e., histopathology (confirmed by the MSKCC Department of Pathology) or BM metastases plus high urine catecholamine levels, or (2) a tumor that is GD2-positive by immunostaining with m3F8.

  °A non-NB tumor is defined as GD2-positive by immunostaining with m3F8. If fresh or frozen tumor is not available for immunostaining, patients will be considered eligible if published reports show that >50% of that tumor type is GD2-positive by immunohistochemistry. (Note: Tissues must be fresh/frozen as fixed, paraffin-embedded specimens are unsuitable for anti-GD2 immunostaining). Tumors known to be GD2-positive by this criteria do not need immunostaining. These include: Melanoma (>50%), Desmoplastic small round cell tumors (70%), Osteosarcoma (88%) and Soft tissue sarcomas including liposarcoma, fibrosarcoma, malignant fibrous histiocytoma, leiomyosarcoma, and spindle cell sarcoma (93%).
* Patients must have either (1) refractory or relapsed high-risk NB (including MYCN-amplified stage 3/4/4S and MYCN-nonamplified stage 4 in patients greater than 18 months of age) resistant to standard therapy, or (2) refractory or relapsed GD2-positive tumor.
* Patients must be older than 1 year of age.
* Prior treatment with murine 3F8 is allowed. Patients with prior m3F8 or ch14.18 treatment must have HAHA antibody titer less than the upper limit of normal [defined as mean + 3*SD of normal volunteers].
* Negative serum pregnancy test in women of childbearing potential.
* Women of child-bearing potential must be willing to practice an effective method of birth control while on treatment
* Signed informed consent indicating awareness of the investigational nature of this program.

Exclusion Criteria:

* Existing major organ dysfunction > grade 2, with the exception of hearing loss and myelosuppression defined as suppression of all types of WBCs, RBCs and platelets). However, the following parameters must be met: white blood cell count ≥1000/ul, absolute (neutrophil count ≥500/ul absolute lymphocyte count ≥500/ul and platelet count ≥ to 25,000/ul
* Active life-threatening infection.
* Pregnant women or women who are breast-feeding.
* Inability to comply with protocol requirements.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-08-15 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dosage (MTD) | 2 years
  At least 3 patients will be studied at each dosage level and dose escalations will only be carried out if 0/3 or < or = to 1/6 patients have dose-limiting toxicity (DLT). At least six patients will be studied at the maximum tolerated dosage (MTD).

SECONDARY OUTCOMES:
pharmacokinetics of hu3F8 | 2 years
  Pharmacokinetics will be measured by serial blood sampling following the iv doses of hu3F8 during cycle 1. Serum hu3F8 will be measured at the following times after infusion of the first hu3F8 infusion during the first cycle: 0, 5 min, 3h, 6-8h, 24h, 48h, 72h, 96, 120h 168h, 216h and 264 h and will also include peak hu3F8 level after infusion for each of the two hu3F8 injections during the first cycle. Peak hu3F8 level at 5 minutes after hu3F8 infusion on days 3 and 5. Pre-treatment and at 5 min after infusion will also be measured for all hu3F8 infusions during all other cycles.
To assess activity of hu3F8 against NB and other GD2-positive tumors. | 2 years
  For neuroblastoma, anti-tumor activity will be measured by INRC.61 For other solid tumors, the response and progression will be evaluated in this study using the Response Evaluation Criteria in Solid Tumors (RECIST) Committee, version 1.1.62
To quantitate pain during hu3F8 treatment | 2 years
  As patient's pain will be assessed with a numerical score of 1 to 10 over the course of the treatment, a curve of pain intensity over time can be generated for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Basu, MD,PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm